CLINICAL TRIAL: NCT06073171
Title: Genomic Study of Cutis Tricolor
Acronym: Cutis Tricolor
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Collaborators: IntegraGen SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RECHMPL22_0229; 2023-A00313-42 (Other: ANSM)
Record Dates: First submitted 2023-05-19; First posted 2023-10-10 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Pigmentary; Dermatosis
MeSH Terms: conditions — Skin Diseases | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cutis Tricolor patient included in trio or duo (Other): Cutis Tricolor patient included in trio (one affected parent, one unaffected parent) or duo (one of the two affected parents)
  Interventions: Biological: Blood sample; Biological: Cutaneous biopsy; Genetic: High troughput sequencing of human's exome

INTERVENTIONS:
Biological: Blood sample — 7.5 mL will be sampled on EDTA tube for each patient
Biological: Cutaneous biopsy — 4 mm of damaged skin will be sampled after a premedication with lidocaine gel for 4 patients
Genetic: High troughput sequencing of human's exome — Sequencing on Illumina NovaSeq6000 platform, using the Twist Bioscience Human Core Exome kit + IntegraGen content, average 37Mb. This sequencing will be realised by external provider, IntegraGen society.

SUMMARY:
It's a study on Syndromic or Isolated Cutis Tricolor and had as main goal to identify the associated gene to the disease thanks to genetic analysis on minors patients and their parents reach by cutis Tricolor or not.

DETAILED DESCRIPTION:
Cutis Tricolor (CT) is a rare cutaneous anomaly defined by pigmentary disorders associating large hyper- and hypopigmented macules of immediate proximity, selectively affecting the trunk. CT can be isolated, sporadic or integrated as a complex syndromic form such as Ruggieri-Happle syndrome (RHS) or various forms of pigmentovascular phacomatosis. A recent analysis of one case of RHS followed by CHU of Montpellier by whole exome sequencing allows the identification of a frameshift pathogen variant (heterozygous state) of a candidate gene.

The main objective is to confirm the association of the candidate gene with syndromic CT (SCT, Ruggierri-Happle syndrome) and non syndromic CT, from a genetic molecular blood and biopsy analysis of patients reach by CT and their parents presenting the disease or not. Furthermore, other objectives are to identify others associated candidates genes and to know better cutaneous pigmentary troubles factors, neurologics and eye abnormalities by identifying the differents cellulars pathways particularly the inflammatory pathway in the pathology of SCT.

First of all, it will have a pre-inclusion visit where Dr WILLEMS. M (Clinical Genetic Department - CHU Montpellier, France) and Pr BESSIS. D (Dermatology Department - CHU Montpellier, France) will explain the study's progress. Then, during the inclusion visit, families will sign inform consent for inclusion in the study. The same day, datas will be collected on demographic, clinical datas, including (i) a description of cutaneous, morphologic and extra-cutaneous anomalies and (ii) a cutaneous biopsy and (iii) a blood test will be done.

The genetics exams results will be return to patients during an usual follow-up visit, 12 months after their inclusion in the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Cutis Tricolor in trio (an affected parent, an unaffected parent) or in duo (one of the two affected parents)
* Age : from 4 to 60 years

Exclusion Criteria:

* Refusal to sign the informed consent
* Patient who doesn't have a social security scheme or beneficiary of such a scheme
* Pregnant or breastfeeding women
* Patient whith a legal protection measure (guardianship, curatorship)
* Patient under legal protection

Ages: 4 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-06-05 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients in whom a pathogenic or probably pathogenic variant has been identified by exome sequencing | 12 months

SECONDARY OUTCOMES:
Number of patients in whom a pathogenic or probably pathogenic variant in the same gene as another patient in the series has been identified | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- University, Montpellier, Montpellier, France